CLINICAL TRIAL: NCT06036433
Title: Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Effectiveness of Photobiomodulation With Exercise, to Enhance Motor, Cognition and the Quality of Life of Those With Parkinson's Disease
Brief Title: Light Therapy Plus Exercise to Improve Motor, Non-Motor Symptoms and QoL in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaitway Neurophysio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBM&exerciseforPDCanada
Record Dates: First submitted 2022-08-30; First posted 2023-09-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's; Disease
Keywords: Photobiomodulation; Light; Laser; Therapy; Transcranial; Abdominal; Neurologic; Neurodegenerative
MeSH Terms: conditions — Parkinson Disease; Disease; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: There are two study arms; the first is a randomized, controlled, double-blind design with Real (Active) and Placebo groups. The study will evaluate the effect of light therapy (photobiomodulation - PBM) on treating the symptoms of moderate-stage PD. Regular exercise is a study prerequisite and must continue throughout the study. There are 30 per group, ages 55-80. Both groups will complete 30-minute, at-home PBM treatments, 3 days/week x 8 weeks (total of 24). Then devices are returned. Subjects have outcome measurement testing at Entry and the end of Weeks 1 & 4 after the last PBM treatment.
  The Crossover includes both the Active & Placebo groups interested in participating in the same 8-week at-home Real PBM protocol outlined above. The same education and weekly support in the first arm is provided in the second arm of the study. Then the devices are returned. Outcome measurement testing will be conducted 1 and 4 weeks after the last PBM treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are unaware of which device they are receiving. The outcomes assessor is unaware of subject randomization and is not involved with any teaching or follow-up of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized, Placebo Controlled, Double-Blind Clinical Trial Real ( Active) vs. Placebo (Sham) (Active Comparator): The first arm includes the real (active) group (n=30) and the placebo (sham) group (n=30). Both groups will self-administer their at-home photobiomodulation (PBM) therapy with devices that either emit active light energy or emit no light energy, respectively. The 30 minute treatment is completed 3 x per week. The protocol includes abdominal PBM treatment with a hand held infrared device and transcranial PBM treatment with an infrared & red LED helmet. Participants are taught how to administer their own treatment and are provided with weekly follow-up. At the completion of the 24 treatments the devices are returned. Post outcome measurement testing is conducted at baseline and 1 and 4 weeks after the last PBM treatment. An inclusion criteria requires that subjects have been exercising 3 x per week before entering the study and continue the minimum level of exercise throughout the study.
  Data from the Real group will be compared with the results from in the Placebo group.
  Interventions: Device: Infrared laser photobiomodulation device; Device: Infrared & Red LED photobiomodulation device
- Active and Placebo Cross Over (Other): After the first arm of the study is completed and the post treatment assessments administered, participants in the Active and Placebo groups will be offered the option to complete 8 weeks of real (active) at-home PBM treatment of the abdomen and head (transcranial), 3 x per week for a total of 24 treatments. Each treatment takes approximately 30 minutes to complete. The devices are then returned. Outcome measurement testing will be conducted at Weeks 1 and 4 weeks after the last treatment.
  Interventions: Device: Infrared laser photobiomodulation device; Device: Infrared & Red LED photobiomodulation device

INTERVENTIONS:
Device: Infrared laser photobiomodulation device — 904 super pulsed Infrared laser PBM therapy for the treatment of the signs and symptoms associated with Parkinson's, such as improved motor, non-motor and Quality of Life.
  Other Names: PDCare Laser by Symbyx Biome Therapies
Device: Infrared & Red LED photobiomodulation device — Infrared & red LED therapy for the treatment of the signs and symptoms associated with Parkinson's, such as motor, non-motor and Quality of Life.
  Other Names: PDNeuro v2.0 by Symbyx

SUMMARY:
Parkinson's disease (PD) is a lifelong and progressive disease and is the second most common progressive neurodegenerative disease worldwide.

This study will examine whether there are significant differences in motor (e.g., balance and gait) and non-motor (e.g., cognition, mood, smell & sleep ) symptoms and quality of life between the Real (active) at-home photobiomodulation (light therapy) combined with exercise group and the Placebo (sham) at-home photobiomodulation (light therapy) combined with exercise group. Each group (Real & Placebo) will include 30 participants; with moderate PD, ages 55-80. Three outcome measurement sessions will be conducted; at the study entry and the end of Weeks 1 & 4 after the last light therapy treatment. Exercise must have been part of the participant's routine before entering the study and will continue during and after the light therapy treatments have been completed.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a lifelong and progressive disease; symptoms slowly worsen over time. PD worldwide is the second most common progressive neurodegenerative disease after Alzheimer's disease. To date there is no cure and few long term effective treatment options.

This research study will use two photobiomodulation (light therapy) devices for at-home treatment by the participant using near-infrared (NIR) and visible red photobiomodulation (PBM). Eligible individuals include those with moderate stage PD and between 55-80 years old. The Real (Active) Group (n=30) will be compared with the Placebo (Sham) group (n=30) to determine whether there are significant differences in motor, cognition and QoL. Exercise will have been part of the subject's routine before entering the study and will continue after the PBM treatments have been completed.

PBM treatments include abdominal and transcranial applications. We believe this is the first combined PBM treatment protocol being used in Canada. Placebo and Real PBM devices look and function the same. The treatment protocol used in this trial is similar to recent Australian PD research using a combination of laser and light-emitting diode (LED) treatments. For almost 20 years, similar transcranial LED parameters have been used safely and effectively to treat traumatic brain injury (TBI), aphasia post stroke and Alzheimer's disease and other dementias.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist-diagnosed Hoehn and Yahr Stages 2-3 (moderate) idiopathic PD;
* With or without anti-Parkinson's Disease medications;
* Able to attend the PD Wellness & Innovation Centre in Hamilton, Ontario, Canada,
* Participating in exercise program prior to enrolment

Exclusion Criteria:

* Previous PBM treatment
* MOCA score of ≤23/30
* Insufficient understanding of English to sign an informed consent, understand teaching and to perform at-home PBM treatment
* Physically unable to perform tasks required for outcome measurement testing
* History of significant unstable musculoskeletal or neurological disorders or unstable cardiac condition

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Timed up-and-go (TUG) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment. (TUG) test | Administered in Arm 1 & 2 at baseline and 1 and 4 weeks after treatment has been completed. Each arm is 12 weeks.
  Time taken to stand from a chair, walk 3m, turn around at a marker, return and sit down. Lower time is a better outcome.

SECONDARY OUTCOMES:
Parts I-VI of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS UPDRS) - to measure change from baseline compared to Endpoints at 1 and 4 weeks Post Treatment | Administered in Arms 1 & 2 at baseline and at Weeks 1 & 4 post treatment. Each arm is 12 weeks.
  Part I) Mentation, Behavior, and Mood, scored in time, range 0-16, lower score is a better outcome; II) ADL score is 0-52, lower score is better outcome: III) Motor portion, score 0-108, lower score is better outcome; IV) Complications of Therapy (in the past week), scores from 0-23, lower is better outcome; V) Modified Hoehn and Yahr Scale, score from 1-5, lower score is better outcome and VI) Schwab and England ADL scale is scored as a percentage, a lower percentage is a better outcome.
10-meter walk Test (10MWT) speed and stride to measure change from baseline compared to Endpoints at weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 weeks.
  assessment of gait, scored by timing completion and counting steps, lower scores are a better outcome.
Montreal Cognitive Assessment (MoCA) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 weeks.
  assessment of cognitive abilities, scored 0-30 (higher scores are better.)
Nine-hole peg test (NHPT) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 weeks.
  test for fine motor skills, timing both the dominant and non-dominant hands. Faster times are a better outcome.
Spiral Test to measure fine motor change from baseline compared with Weeks 1 & 4 post treatment. | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 weeks.
  Spiral drawing is a skilled and complex coordinated motor activity. Scores are based on time and accuracy, a lower scores is a better outcome.
Writing Test to measure fine motor changes from baseline compared to Weeks 1 & 4 post treatment. | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 weeks in duration.
  Writing test is administered to assess for bradykinesia, micrographia and tremor in Parkinson's disease. Size and quality of writing determine outcome or change.
Parkinson's Disease Quality of Life 39 (PDQ39) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 4 post treatment. Each arm is 12 week. .
  Quality of Life, scored in percentage (0-100%), lower score is a better outcome.
Parkinson's Disease Sleep Scale ( PDSS) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 2 post treatment. Each arm is 12 weeks.
  self-rate and quantify the level of sleep disruption, 0-60, lower score is a better outcome.
Smell test to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 2 post treatment. Each arm is 12 weeks.
  Investigator administers 4 scents to evaluate the sense of smell, scored between 0-12; higher score is a better outcome.
Beck Depression Inventory (BDI) to measure change form baseline compared to Endpoints at Weeks 1 and 4 post treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 2 post treatment. Each arm is a total of 12 weeks in total.
  is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression; lower score is a better outcome.
Beck Anxiety Inventory (BAI) to measure change from baseline compared to Endpoints at Weeks 1 and 4 Post Treatment | Administered in Arms 1 & 2 at baseline and Weeks 1 & 2 post treatment. Each arm is a total of 12 weeks.
  is a 21-question multiple-choice self-report inventory used to measure how the subject has been feeling in the last week, focusing primarily on somatic symptoms; lower score is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Saltmarche, MHSc, Study Chair — Saltmarche Health & Associates; Orla Hares, PT, Principal Investigator — Neuro Physio at Gaitway Neurophysio and Parkinson's Wellness Innovation Centre
Locations (1):
- Gaitway Neurophysio and Parkinson's Wellness Innovation Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study is being conducted at Parkinson's Wellness & Innovation Centre — https://gaitwayneurophysio.com/